CLINICAL TRIAL: NCT03733119
Title: ONC201 With a Methionine-Restricted Diet in Patients With Metastatic Triple Negative Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: The V Foundation for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW17107; 2018-0252 (Other: Institutional Review Board); A534260 (Other: UW Madison); SMPH/MEDICINE/HEM-ONC (Other: UW Madison); NCI-2018-01878 (Registry Identifier: NCI Trial ID); Protocol Version 02/16/2021 (Other: UW Madison)
Record Dates: First submitted 2018-11-05; First posted 2018-11-07 (Actual); Results first posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — TIC10 compound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Akt/ERK inhibitor ONC201 (Experimental): Participants receive Akt/ERK inhibitor ONC201 PO on days 3, 10, and 17. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Akt/ERK Inhibitor ONC201
- Akt/ERK inhibitor ONC201, methionine-restricted diet (Experimental): Participants receive Akt/ERK inhibitor ONC201 PO on days 3, 10, and 17. Participants also receive methionine-restricted diet PO on days 1-5, 8-12, and 15-19. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Akt/ERK Inhibitor ONC201; Dietary Supplement: Methionine-Restricted Diet

INTERVENTIONS:
Drug: Akt/ERK Inhibitor ONC201 — Given PO
  Other Names: ONC201; TIC10
Dietary Supplement: Methionine-Restricted Diet — Given PO
  Arms: Akt/ERK inhibitor ONC201, methionine-restricted diet

SUMMARY:
This phase II trial studies how well Akt/ERK inhibitor ONC201 (ONC201) with a methionine-restricted (MR) diet works in treating participants with triple negative breast cancer that has spread to other places in the body or cannot be removed by surgery. ONC201 activates a process that leads to the death of a cell. ONC201 is able to target tumor cells to get rid of them, but does not affect normal cells. MR diet is a methionine-free amino acid modified medical food. The addition of an intermittent MR diet may enhance the activity of ONC201. Giving ONC201 and an MR diet may work better in treating participants with breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine objective response rate (ORR) to ONC201 with a methionine-restricted diet in patients with metastatic triple negative breast cancer (TNBC).

SECONDARY OBJECTIVES:

I. To determine progression-free survival (PFS) to ONC201 with a methionine-restricted diet in patients with metastatic TNBC.

II. To determine clinical benefit rate (complete or partial response plus stable disease) (CBR) at 4 months to ONC201 with a methionine-restricted diet in patients with metastatic TNBC.

III. To determine overall survival (OS) to ONC201 with a methionine-restricted diet in patients with metastatic TNBC.

IV. To assess metabolic indices in patients with metastatic TNBC treated with ONC201 and a methionine-restricted diet.

V. To assess the expression of TRAIL receptor in circulating tumor cells (CTCs) prior, during and upon progression in patients with metastatic TNBC treated with ONC201 with a methionine-restricted diet.

EXPLORATORY OBJECTIVES:

I. To determine time to development of brain metastases or worsening of brain metastases in patients with metastatic TNBC treated with ONC201 with a methionine-restricted diet.

STUDY DESIGN Patients with metastatic TNBC will be enrolled in a single-arm study evaluating ONC201 with a methionine-restricted diet.

After completion of study treatment, participants are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic or unresectable TNBC (estrogen receptor [ER] < 10%, progesterone receptor [PR] < 10% and HER2 negative either by immunohistochemistry [IHC] or in situ hybridization method by American Society of Clinical Oncology [ASCO]-College of American Pathologists [CAP] guidelines). For patients with a previous tumor sample with positive ER, PR and/or HER2 results, if the most recent biopsy meets study criteria, they will be eligible.
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. within 28 days prior to registration
* Written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately
* Any number of prior lines of systemic therapy for metastatic disease
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
* Prior cancer treatment, including radiotherapy, must be completed at least 14 days prior to registration and the subject must have recovered from all reversible acute toxic effects of the regimen to =< grade 1 or to baseline prior to initiation of that therapy. Grade 2 or higher exceptions include alopecia, up to grade 2 neuropathy, and other grade 2 AEs or lab values not constituting a safety risk in the opinion of the treating physician. This criteria does not apply to lab tests for normal organ and marrow function outlined below.
* No active central nervous system (CNS) metastatic disease; subjects with prior definitive treatment of their CNS disease by surgical resection, stereotactic body radiation therapy (SBRT) or whole-brain radiotherapy (WBRT) > 28 days ago will be eligible if asymptomatic and off systemic steroids
* Life expectancy of greater than 12 weeks
* Normal organ and marrow function as defined per protocol definitions

  * Absolute neutrophil count (ANC) > 1.5 x 10^3/uL
  * Platelet count >= 100 x 10^3/uL
  * Hemoglobin >= 9 g/dL
  * Total bilirubin < 1.5 x upper limit of normal (ULN)
  * Aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT)/serum glutamic-pyruvic transaminase (SGPT) ≤ 2.5 x ULN if participant has liver metastases, ≤5x ULN.
  * Creatinine < ULN (institutional normal)
* Females of childbearing potential must have a negative serum pregnancy test within 7 days prior to registration. NOTE: Females are considered of childbearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy), or they are naturally postmenopausal for at least 12 consecutive months
* Females of childbearing potential must be willing to abstain from heterosexual activity or must agree to use adequate contraception (hormonal or barrier method) for the duration of study participation and for 90 days after discontinuation of study treatment
* Ability of the subject to understand and comply with study procedures for the entire length of the study
* Able to swallow ONC201
* Be willing to discontinue vitamin and mineral supplements for the duration of the study if randomized to receive the methionine restricted diet

Exclusion Criteria:

* No prior therapy with TRAIL receptor agonists
* Active infection requiring systemic therapy. Patients with a known history of human immunodeficiency virus (HIV) must have a CD4 count >= the institutional lower limit of normal within 28 days prior to registration. Patients with HIV must also be on a stable antiretroviral regimen for >= 28 days before registration
* Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study)
* Known additional malignancy that is active and/or progressive requiring treatment; exceptions include basal cell or squamous cell skin cancer, in situ cervical or bladder cancer, or other cancer for which the subject has been disease-free for at least three years
* Treatment with any investigational drug agent =< 14 days prior to registration or within 5 half-lives of that investigational product, whichever is longer
* Participant who has had major surgery =< 14 days prior to registration or has not recovered from major side effects of the surgery (tumor biopsy is not considered as major surgery)
* Known hypersensitivity to any of the excipients of ONC201
* Any impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* Any concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, cause unacceptable safety risks, contraindicate subject participation in the clinical study or compromise compliance with the protocol (e.g. chronic pancreatitis, chronic active hepatitis, active untreated or uncontrolled fungal, bacterial or viral infections, etc.)
* Participants who follow a vegan or vegetarian diet

Ages: 18 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2021-02-13 (Actual); Study Completion 2021-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kari Wisinski, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liao M, Qin R, Huang W, Zhu HP, Peng F, Han B, Liu B. Targeting regulated cell death (RCD) with small-molecule compounds in triple-negative breast cancer: a revisited perspective from molecular mechanisms to targeted therapies. J Hematol Oncol. 2022 Apr 12;15(1):44. doi: 10.1186/s13045-022-01260-0. PMID 35414025
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 4 participants enrolled, 1 determined not to meet the eligibility criteria, 3 participants started treatment
Period: Overall Study
Arm/Group | Akt/ERK Inhibitor ONC201 | Akt/ERK Inhibitor ONC201, Methionine-restricted Diet
Started | 2 | 2
Treated | 2 | 1
Stopped Treatment After 1 Dose (removed by physician for disease progression 2 days after first dose) | 1 | 0
Stopped Treatment After 3 Cycles (removed by physician for disease progression after the first planned time point for disease evaluation) | 1 | 1
Completed | 0 | 0
Not Completed | 2 | 2
Not completed — Physician Decision | 2 | 1
Not completed — ineligible to treat per protocol | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Akt/ERK Inhibitor ONC201 | Akt/ERK Inhibitor ONC201, Methionine-restricted Diet | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Customized [Count of Participants; unit: Participants]
  Age (years): 20-29 | 0 | 1 | 1
  Age (years): 30-39 | 0 | 0 | 0
  Age (years): 40-49 | 1 | 0 | 1
  Age (years): 50-59 | 1 | 0 | 1
  Age (years): 60-69 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) - Number of Participants Who Responded to Treatment
Description: ORR will be estimated according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, by dividing the total number of responders (complete plus partial responses plus CR or PR) or (CR or PR), respectively, by number of subjects with measurable disease and the exact 95% confidence interval will be provided.
  Due to early termination with few participants, only the counts of events have been reported.
Time Frame: maximum follow up time was 1 year
Population: study was terminated early, data for response rate at 2 years per protocol was not collected
Measure: Count of Participants; unit: Participants
Arm/Group | Akt/ERK Inhibitor ONC201 | Akt/ERK Inhibitor ONC201, Methionine-restricted Diet
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0

2. Secondary Outcome: Progression-free Survival (PFS) - Number of Participants With PFS
Description: Will be summarized using Kaplan-Meier estimates of the median survival times. Point estimates as well as 95% confidence intervals will be provided.
  Due to early termination with few participants, only the counts of events have been reported.
Time Frame: maximum follow up time was 1 year
Population: study was terminated early, data for progression free survival at 2 years not collected
Measure: Count of Participants; unit: Participants
Arm/Group | Akt/ERK Inhibitor ONC201 | Akt/ERK Inhibitor ONC201, Methionine-restricted Diet
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0

3. Secondary Outcome: Overall Survival (OS) - Number of Participants Who Survived the Study Period
Description: as for outcome 2
Time Frame: maximum follow up time was 1 year
Population: study was terminated early, data for overall survival at 2 years not collected
Measure: Count of Participants; unit: Participants
Arm/Group | Akt/ERK Inhibitor ONC201 | Akt/ERK Inhibitor ONC201, Methionine-restricted Diet
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0

4. Secondary Outcome: Clinical Benefit Rate (CBR) - Number of Participants Who Experienced Clinical Benefit
Description: CBR will be estimated according to RECIST 1.1, by dividing the total number of responders (complete plus partial responses plus CR or PR or stable disease [SD]), by number of subjects with measurable disease and the exact 95% confidence interval will be provided.
  Due to early termination with few participants, only the counts of events have been reported.
Time Frame: At 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Akt/ERK Inhibitor ONC201 | Akt/ERK Inhibitor ONC201, Methionine-restricted Diet
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0

5. Secondary Outcome: Duration of Response (DOR)
Description: Will be measured using Kaplan-Meier methodology. A 95% confidence interval will be provided for the median duration of response.
Time Frame: Up to 2 years
Population: duration of response could not be calculated as there were no responders on study
Arm/Group | Akt/ERK Inhibitor ONC201 | Akt/ERK Inhibitor ONC201, Methionine-restricted Diet
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Incidence of Adverse Events - Number of Participants Who Experienced Adverse Events
Description: Incidence of adverse events as measured by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) 5.0. Safety and tolerability will be assessed by frequency tables. Also, metabolic indices in patients with metastatic triple negative breast cancer (TNBC) treated with ONC-201 and a methionine-restricted diet will be assessed by frequency tables and descriptive statistics.
Time Frame: 30 days after last dose of study drug, up to 4 months on study
Population: See Adverse Events Module for a complete summary of adverse events data.
Measure: Count of Participants; unit: Participants
Arm/Group | Akt/ERK Inhibitor ONC201 | Akt/ERK Inhibitor ONC201, Methionine-restricted Diet
Number analyzed (Participants) | 2 | 1
Participants | 2 | 1

7. Other Pre Specified Outcome: Time to Development or Worsening of Brain Metastases
Description: Will be summarized using Kaplan-Meier methodology.
Time Frame: Up to 2 years
Population: study was terminated early, data for outcome at 2 years not collected, see Number of Participants with Development or Worsening of Brain Metastases Outcome for more information
Arm/Group | Akt/ERK Inhibitor ONC201 | Akt/ERK Inhibitor ONC201, Methionine-restricted Diet
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Number of Participants With Developing or Worsening Brain Metastasis
Time Frame: up to 4 months
Population: one participant was determined to have a brain metastasis prior to treatment, outcome measure added to provide additional information about participant population
Measure: Count of Participants; unit: Participants
Arm/Group | Akt/ERK Inhibitor ONC201 | Akt/ERK Inhibitor ONC201, Methionine-restricted Diet
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 4 months
Description: Participants were followed for 30 days after last dose of study drug
Arm/Group | Akt/ERK Inhibitor ONC201 | Akt/ERK Inhibitor ONC201, Methionine-restricted Diet
All-Cause Mortality (participants affected / at risk) | 2/2 | 1/1
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Akt/ERK Inhibitor ONC201 (N=2) | Akt/ERK Inhibitor ONC201, Methionine-restricted Diet (N=1)
Pericardial tamponade (Cardiac disorders) | 1 (1) | 0 (0) — Reported as an SAE - event occurred more than 30 days post treatment and was determined to be disease related.
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) — Reported as an SAE - event occurred more than 30 days post treatment and was determined to be disease related.
Lung infection (Infections and infestations) | 1 (1) | 0 (0) — Reported as an SAE - event occurred more than 30 days post treatment and was determined to be disease related.
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Akt/ERK Inhibitor ONC201 (N=2) | Akt/ERK Inhibitor ONC201, Methionine-restricted Diet (N=1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnea (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (1)
Fever (General disorders) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Hemoglobinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 1 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (2)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vision decreased (Eye disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (4) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 1 (2)

LIMITATIONS AND CAVEATS:
Trial was terminated early due to slow accrual, not powered for meaningful results, statistical analysis not completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/19/NCT03733119/Prot_SAP_000.pdf